CLINICAL TRIAL: NCT04823247
Title: A Multicenter, Prospective Observational RWE Study to Assess Patient-reported Wellbeing Using Tildrakizumab in a Live Setting - POSITIVE Study
Brief Title: Observational Real-world Evidence (RWE) Study to Assess Patient-reported Wellbeing Using Tildrakizumab in Live Setting - POSITIVE Study
Acronym: POSITIVE
Status: Completed | Type: Observational
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: M-14745-47
Record Dates: First submitted 2021-03-24; First posted 2021-03-30 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Plaque Psoriasis
Keywords: Moderate-to-severe plaque psoriasis; Psoriasis; Tildrakizumab; Prospective
MeSH Terms: conditions — Psoriasis | interventions — tildrakizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tildrakizumab: Patients diagnosed with moderate-to-severe plaque psoriasis who require systemic biologic therapy and qualify for treatment with an IL-23p19 inhibitor in real-world clinical practice, following the routine clinical practice on each patient country, will be observed for 24 months.
  Interventions: Drug: Tildrakizumab

INTERVENTIONS:
Drug: Tildrakizumab — As provided in real world clinical practice.
  Other Names: IL-23p19 inhibitor

SUMMARY:
This is an ethics-approved, multi-national, multi-site Phase IV, 1-cohort prospective observational study. The main purpose of this study is to assess the effect of tildrakizumab on the overall wellbeing in patients with moderate-to-severe psoriasis using the 5-item World Health Organization Wellbeing Index (WHO-5) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosis of moderate-to-severe chronic plaque psoriasis documented in the medical chart.
* Patient who need systemic biologic therapy and qualify for treatment with an IL-23p19 inhibitor. Tildrakizumab must be the anti-IL-23p19 selected therapy before including the patient in the study.
* Patient aged 18 years or older at the time of patient recruitment.
* Patient who have provided written informed consent (if required by country regulations).

Exclusion Criteria:

* Patients unable to comply with the requirements of the study (fulfilling of the study questionnaires) or who, in the opinion of the study physician, should not participate in the study.
* Patients included in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with moderate-to-severe plaque psoriasis who need systemic biologic therapy and qualify for treatment with an IL-23p19 inhibitor treatment in real-world clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 782 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in 5-item World Health Organization Wellbeing Index (WHO-5) Score | Baseline and Month 24

SECONDARY OUTCOMES:
Change From Baseline in 5-item World Health Organization Wellbeing Index (WHO-5) Score | Baseline; 16 and 28 weeks; 12, 18 months after baseline visit
Change from Baseline in Physician's Satisfaction Questionnaire Score | Baseline; 16 and 28 weeks; 12, 18 and 24 months after baseline visit
Change from Baseline in FamilyPso Questionnaire Score | Baseline; 16 and 28 weeks; 12, 18 and 24 months after baseline visit
Change From Baseline in Dermatology Life Quality Index-Relevant (DLQI-R) Score | Baseline; 16 and 28 weeks; 12, 18 and 24 months after baseline visit
Change From Baseline in Treatment Satisfaction Questionnaire for Medication (TSQM-9) Score | Baseline; 16 and 28 weeks; 12, 18 and 24 months after baseline visit
Change From Baseline in Treatment-related Patient Benefit Index 2.0 (PBI 2.0) Score | Baseline; 16 and 28 weeks; 12, 18 and 24 months after baseline visit
Change From Baseline in Work Productivity and Activity Impairment Questionnaire: Psoriasis (WPAI:PSO) Score | Baseline; 16 and 28 weeks; 12, 18 and 24 months after baseline visit
Skin Manifestations Distribution (Patient's Grid/Heat Map) | Baseline; 16 and 28 weeks; 12, 18 and 24 months after baseline visit
Change from Baseline in Numerical Rating Scale (NRS) Scores for Itch, Pain, Joint Pain and Fatigue | Baseline; 16 and 28 weeks; 12, 18 and 24 months after baseline visit
Change from Baseline in Psoriasis Area and Severity Index (PASI) Score | Baseline; 16 and 28 weeks; 12, 18 and 24 months after baseline visit
Number of Patients Compliance to Sociodemographic Characteristics and Clinical Characteristics | From Baseline up to 24 months
Number of Patients With Treatment-emergent Adverse Events (TEAE) | From Baseline up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Haut- und Laserzentrum Freising, Freising, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mrowietz U, Sommer R, Gerdes S, Reguiai Z, Weger W, Dauden E, Maul JT, Ghislain PD, Laws PM, Naldi L, De Jong E, Mburu S, Koscielny V, Massana E, Domenech A, Gaarn du Jardin K, Kasujee I, Augustin M. Patient-Reported Well-Being in Value-Based Routine Care Using Tildrakizumab: 52-week Interim Data of the Phase IV Positive Study. Psoriasis (Auckl). 2025 Jun 28;15:243-259. doi: 10.2147/PTT.S526748. eCollection 2025. PMID 40605963
- [Derived] Augustin M, Sommer R, Dauden E, Laws P, de Jong E, Fabbrocini G, Naldi L, Navarini A, Lambert J, Reguiai Z, Gerdes S, Massana E, Obis T, Kasujee I, Mrowietz U. Patient-reported well-being in value-based care using tildrakizumab in a real-world setting: protocol of a multinational, phase IV, 1-cohort prospective observational study (the POSITIVE study). BMJ Open. 2023 Feb 15;13(2):e060536. doi: 10.1136/bmjopen-2021-060536. PMID 36792337